CLINICAL TRIAL: NCT06718309
Title: A Prospective Cohort Study of Chemotherapy Plus Immunotherapy Combined With Stereotactic Body Radiotherapy as Neoadjuvant Therapy for Patients With Resectable Non-small Cell Lung Cancer
Brief Title: Chemotherapy Plus Immunotherapy Combined With SBRT as Neoadjuvant Therapy for Patients With Resectable NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZCH-2024-003
Record Dates: First submitted 2024-11-24; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; locally advanced; resectable; SBRT; immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Immunotherapy

STUDY DESIGN:
Intervention Model Description: In this study, patients with surgically resectable locally advanced non-small cell lung cancer (stage II-IIIA and part of stage IIIB) (EGFR/ALK wild-type for adenocarcinoma patients) are enrolled. Eligible patients firstly receive one cycle of chemoimmunotherapy, followed by stereotactic body radiotherapy (SBRT) (8Gy*3F) to the primary lung lesion and then continued with another two cycles of chemoimmunotherapy. Surgical treatment was performed within 4-6 weeks after the last chemoimmunotherapy. Immunotherapy continues until 1 year after surgery. Minimal residue lesion (MRD) are monitored at 5 timepoints during the treatment period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Treatment group
  Interventions: Drug: Chemotherapy; Drug: Immunotherapy; Procedure: Radical resection of lung cancer; Radiation: SBRT

INTERVENTIONS:
Drug: Chemotherapy — Patients with squamous cell carcinoma can choose paclitaxel + cisplatin/carboplatin and patients with nonsquamous cell carcinoma can choose pemetrexed + cisplatin/carboplatin. The chemotherapy treatment lasts 3 cycles.
Drug: Immunotherapy — Investigators choose PD-1 or PD-L1 according to drug indication and the immunotherapy lasts 3 cycles preoperatively and 1 year after surgery.
Procedure: Radical resection of lung cancer — Radical resection of lung cancer with lymph node dissection
Radiation: SBRT — SBRT for primary lung lesion 8Gy*3F after first cycle of chemoimmunotherapy

SUMMARY:
In this study, patients with EGFR/ALK wild-type, resectable locally advanced NSCLC are expected to receive 1 cycle of chemoimmunotherapy as neoadjuvant therapy, followed by SBRT to the primary lung lesion, and chemoimmunotherapy for 2 cycles. Surgical treatment will be given within 4-6 weeks after the last cycle of chemoimmunotherapy, then immunotherapy maintenance for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or pathologically confirmed, newly diagnosed non-small cell lung cancer patients;
2. Age ≥18 years;
3. (Eastern Cooperative Oncology Group, ECOG) (Performance Status, PS) score 0-1;
4. According to the 8th-9th edition of (American Joint Committee on Cancer, AJCC) (stage II-IIIA, for stage IIIB included T3-4N2, T4 only included tumor > 7cm);
5. Puncture or biopsy samples were tested EGFR/ALK negative;
6. Surgically or potentially resectable after discussion by multidisciplinary team (MDT);
7. Who has not received systemic antitumor therapy and has not received chest radiotherapy;
8. Evaluable lesions in the lung or mediastinum;
9. The organ function level should meet the following criteria one week before enrollment: 1) Bone marrow function: hemoglobin ≥80g/L, white blood cell count ≥4.0*10^9/L or neutrophil count ≥1.5*10^9/L, platelet count ≥100*10^9/L; 2) Liver: total serum bilirubin level ≤1.5 times the normal upper limit, when serum total bilirubin level > 1.5 times the normal upper limit, direct bilirubin level ≤ normal upper limit, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 times the normal upper limit; 3) Kidney: blood creatinine level < 1.5 times the normal upper limit or creatinine clearance ≥50ml/min, urea nitrogen ≤200mg/L; Serum albumin ≥30g/L;
10. Male/female of childbearing age agrees to use contraception during the trial period (surgical ligation or oral contraceptives/IUDs + condom contraception);
11. Sign informed consent.

Exclusion Criteria:

1. Patients with severe dysfunctions of the heart, lungs and other organs who are not suitable for surgery;
2. Patients with severe autoimmune diseases: active inflammatory bowel disease (including Crohn's disease, ulcerative colitis), rheumatoid arthritis, scleroderma, systemic lupus erythematosus, autoimmune vasculitis (such as Wegener's granuloma), etc;
3. Other malignancies within 5 years (excluding non-melanoma skin cancer and cervical cancer);
4. Patient with active infection, heart failure, heart attack, unstable angina pectoris or unstable arrhythmia within the last 6 months;
5. Congenital or acquired immunodeficiency disorders include human immunodeficiency virus (HIV) or a history of organ transplantation or allogeneic stem cell transplantation;
6. Patients treated with other immunological agents, chemotherapy agents, other drugs in clinical trials and long-term cortisol therapy were excluded;
7. Patients who are allergic or contraindicated to PD-1 inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | Assessed up to 24 weeks
  Pathological complete response for surgical patients

SECONDARY OUTCOMES:
Major pathologic response (MPR) | Assessed up to 24 weeks
  No more than 10% residual viable tumour in the resected tumour (up to 24 weeks)
1-year event-free survival (1 year EFS) | Assessed up to 100 months
  Interval between the start of neoadjuvant treatment and any progression of disease precluding surgical resection, progression of disease in the absence of surgery, progression or recurrence after surgery, or death from any cause, whichever occurred first
The R0 resection rate | Assessed up to 24 weeks
  The proportion of patients who had complete surgical resection [R0]
Incidence of treatment-related adverse events | assessed up to 100 months
  The incidence of adverse events ≥ grade 3 during perioperative period

CONTACTS AND LOCATIONS:
Overall Officials: Lucheng Zhu, MD, Principal Investigator — Hangzhou Cancer Hospital
Locations (1):
- Department of Thoracic Oncology, Hangzhou Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang JT, Liu SY, Gao W, Liu SM, Yan HH, Ji L, Chen Y, Gong Y, Lu HL, Lin JT, Yin K, Jiang BY, Nie Q, Liao RQ, Dong S, Guan Y, Dai P, Zhang XC, Yang JJ, Tu HY, Xia X, Yi X, Zhou Q, Zhong WZ, Yang XN, Wu YL. Longitudinal Undetectable Molecular Residual Disease Defines Potentially Cured Population in Localized Non-Small Cell Lung Cancer. Cancer Discov. 2022 Jul 6;12(7):1690-1701. doi: 10.1158/2159-8290.CD-21-1486. PMID 35543554
- [Result] Xia L, Mei J, Kang R, Deng S, Chen Y, Yang Y, Feng G, Deng Y, Gan F, Lin Y, Pu Q, Ma L, Lin F, Yuan Y, Hu Y, Guo C, Liao H, Liu C, Zhu Y, Wang W, Liu Z, Xu Y, Li K, Li C, Li Q, He J, Chen W, Zhang X, Kou Y, Wang Y, Wu Z, Che G, Chen L, Liu L. Perioperative ctDNA-Based Molecular Residual Disease Detection for Non-Small Cell Lung Cancer: A Prospective Multicenter Cohort Study (LUNGCA-1). Clin Cancer Res. 2022 Aug 2;28(15):3308-3317. doi: 10.1158/1078-0432.CCR-21-3044. PMID 34844976
- [Result] Qiu B, Guo W, Zhang F, Lv F, Ji Y, Peng Y, Chen X, Bao H, Xu Y, Shao Y, Tan F, Xue Q, Gao S, He J. Dynamic recurrence risk and adjuvant chemotherapy benefit prediction by ctDNA in resected NSCLC. Nat Commun. 2021 Nov 19;12(1):6770. doi: 10.1038/s41467-021-27022-z. PMID 34799585
- [Result] Galluzzi L, Aryankalayil MJ, Coleman CN, Formenti SC. Emerging evidence for adapting radiotherapy to immunotherapy. Nat Rev Clin Oncol. 2023 Aug;20(8):543-557. doi: 10.1038/s41571-023-00782-x. Epub 2023 Jun 6. PMID 37280366
- [Result] Wakelee H, Liberman M, Kato T, Tsuboi M, Lee SH, Gao S, Chen KN, Dooms C, Majem M, Eigendorff E, Martinengo GL, Bylicki O, Rodriguez-Abreu D, Chaft JE, Novello S, Yang J, Keller SM, Samkari A, Spicer JD; KEYNOTE-671 Investigators. Perioperative Pembrolizumab for Early-Stage Non-Small-Cell Lung Cancer. N Engl J Med. 2023 Aug 10;389(6):491-503. doi: 10.1056/NEJMoa2302983. Epub 2023 Jun 3. PMID 37272513